CLINICAL TRIAL: NCT03679312
Title: The Effect of Inhaled Nitric Oxide on Dyspnea and Exercise Tolerance in COPD
Acronym: iNO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University Hospital Foundation (Other); Canadian Lung Association (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00078715
Record Dates: First submitted 2018-09-06; First posted 2018-09-20 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Randomized double-blind cross-over design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COPD Group (Experimental): COPD to receive either placebo or inhaled nitric oxide (40ppm)
  Interventions: Drug: Nitric Oxide; Drug: Placebo
- Control Group (Experimental): Control group to receive either placebo or inhaled nitric oxide (40ppm)
  Interventions: Drug: Nitric Oxide; Drug: Placebo

INTERVENTIONS:
Drug: Nitric Oxide — Inhaled nitric oxide, which consists of breathing medical grade air (21% O2) with 40 parts per million of nitric oxide.
  Other Names: Inhaled Nitric Oxide
Drug: Placebo — Inhaled placebo, which consists of breathing medical grade air (21% O2).
  Other Names: Medical Grade Room Air

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a lung disorder commonly caused by smoking, which makes breathing more difficult. When COPD patients exercise, they are not efficient breathers and this leads to serious breathing difficulties, which often causes these patients to stop exercise at low intensities. Even though patients with a mild form of COPD have relatively well preserved lung function, they still have inefficient breathing during exercise. The investigators think that these patients have problems exchanging fresh gas (i.e., oxygen) into the blood stream because of poor lung blood vessel function. The investigators will test whether inhaled medications, specifically nitric oxide, can improve lung blood vessel function and decrease breathing difficulties during exercise. With this research, the investigators will understand more about breathing efficiency and lung blood vessel function in patients with COPD, and find out whether improving lung blood vessel function helps COPD patients breathe easier and exercise longer. Understanding the reasons behind the feeling of difficult breathing may lead to more effective therapy and improved quality of life in COPD patients.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a respiratory disorder typically caused by smoking and is characterized by airway obstruction. Exertional dyspnea (perceived breathlessness) is a hallmark of COPD regardless of severity and is the primary reason for exercise intolerance even in patients with mild COPD (defined using spirometric criteria as a forced expiratory volume in 1 s (FEV1)/forced vital capacity (FVC) <0.70 and a FEV1 ≥ 80%). Dyspnea in COPD has been shown to profoundly reduce patient quality of life, physical activity, and impair patients' ability to complete day-to-day tasks. Previous work in mild COPD has demonstrated that exertional dyspnea is the result of increased work of breathing during exercise, and that this increased work of breathing comes from: 1) an exaggerated ventilatory response to exercise (i.e. increased minute ventilation relative to carbon dioxide production, V̇E/V̇CO2), and 2) airflow limitation (i.e. expiratory flow limitation and resulting dynamic hyperinflation). A great deal of work has focused on improving airflow limitation in COPD; however, very little has been done to understand and treat the exaggerated ventilatory response to exercise in COPD.

Several previous studies in COPD have consistently shown an elevated ventilatory response (i.e. greater V̇E/V̇CO2) during exercise. The elevated V̇E/V̇CO2 response to exercise appears to be clinically important, as it independently predicts mortality in COPD and indicates that physiological abnormalities beyond airflow obstruction are important in determining disease severity, dyspnea, and risk of death. This increased V̇E/V̇CO2 in COPD appears to be secondary to increased deadspace ventilation(i.e. sections of the lung with ventilation, but no perfusion), and this increased deadspace ventilation results in a compensatory increase in total minute ventilation (i.e. increased V̇E/V̇CO2) to maintain effective alveolar ventilation and arterial blood gas homeostasis.

The underlying mechanism(s) for the increased deadspace ventilation and V̇E/V̇CO2 during exercise in mild to moderate COPD is currently unclear; however, pulmonary microvascular abnormalities and hypoperfusion of pulmonary capillaries are potential pathophysiologic mechanisms. Mild to moderate COPD patients have reduced pulmonary microvascular blood flow in nonemphysematous lung regions, which has led researchers to conclude that the low pulmonary perfusion in an intact pulmonary vascular bed is likely the result of pulmonary vascular dysfunction. Ventilation-perfusion (V̇A/Q̇) data in mild and moderate COPD shows substantial V̇A/Q̇ inequality at rest, with the V̇A/Q̇ distribution skewed towards regions of high V̇A/Q̇, which is indicative of increased deadspace. Consistent with this capillary hypoperfusion hypothesis, our recent work has shown a blunted pulmonary capillary blood volume response to exercise in mild COPD, when compared to age- and height-matched non-smoking controls. Importantly, the low pulmonary capillary blood volume was associated with increased V̇E/V̇CO2 during exercise, suggesting that low pulmonary perfusion (i.e. reduced pulmonary capillary blood volume) leads to increased deadspace.

Inhaled nitric oxide (NO) is commonly used to test for pulmonary vasodilatory responses in patients with pulmonary arterial hypertension (PAH), as it increases NO bioavailability and improves pulmonary vascular function. Previous work in PAH and heart failure (HF) patients has shown that standard doses (20-40 parts per million (ppm)) of inhaled NO can reduce pulmonary vascular resistance and increase peak oxygen consumption (V̇O2peak). If inhaled NO can reduce vascular dysfunction and increase perfusion in mild and moderate COPD, this would result in a reduction in V̇E/V̇CO2 and improved exercise tolerance.

STUDY PURPOSE

Purpose: To examine the effect of inhaled NO on exercise capacity (V̇O2peak) ventilation and dyspnea in in patents with COPD.

Hypothesis: Inhaled NO will improve exercise capacity, secondary to reduced V̇E/V̇CO2 and dyspnea, in mild and moderate COPD, while no change will be observed in healthy controls and severe COPD.

Study Design: Randomized double-blind cross-over design.

All participants will have a pulmonary function and cardiopulmonary exercise test. The study procedure is briefly outlined below and is further outlined in the attached University Hospital Foundation Grant.

Study Protocol: Seven sessions will be completed over a 3-week period in the following order:

Day 1) Participant enrollment, medical history, standard pulmonary function (PFT) and cardiopulmonary exercise test (CPET).

Days 2 & 3) Randomly-ordered experimental CPETs while either breathing room air or inhaled nitric oxide (room air with 40 ppm NO).

Days 4 & 5) Randomly-ordered constant load exercise tests, at 75% peak power output, while either breathing room air or inhaled nitric oxide (room air with 40 ppm NO).

Day 6) Ultrasonography doppler measurements will be completed to determine pulmonary arterial systolic pressure (at rest and during exercise) while breathing room air or inhaled nitric oxide. Doppler measurements of systemic vascular endothelial function will be measured at rest while breathing room air. To enhance doppler signal during the cardiac ultrasound, agitated saline contrast will be used. A small sample of venous blood will be taken to analyze inflammatory levels. Additionally, participants will breathe into a small tube so that expelled saliva can be analyzed to determine airway inflammation.

Day 7) Prospective quantitative computed tomography (CT) imaging will be completed to obtain lung density, heterogeneity, tissue, vascular and airway measurements.

Each visit will take approximately 3 hours. The total time duration for each participant will be approximately 21 hours.

ELIGIBILITY:
Inclusion Criteria - COPD Patients:

* No significant cardiovascular disease.
* No significant metabolic disease
* No significant neuromuscular disease
* Participants will range from 18-85 years old

Inclusion Criteria - Control Patients:

* Age- and sex-matched to COPD patients
* Normal lung function
* Minimal smoking history
* No previous diagnosis of COPD
* Participants will range from 18-85 years old

Exclusion Criteria:

* Individuals with significant cardiovascular, metabolic, neuromuscular or any other disease
* Individual with musculoskeletal injuries
* Individuals currently on oral steroids (i.e. prednisone), phosphodiesterase type 5 (PDE5) inhibitors or supplemental O2 therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Peak Workload | Within 20-25 minutes post-dose
  Peak workload will be defined as the highest wattage obtained during a 20 s period during the test.
Peak Oxygen Consumption | Within 20-25 minutes post-dose
  Peak oxygen consumption will be defined as the highest O2 uptake (reported in ml/kg/min) obtained during a 20 s period during the test.

SECONDARY OUTCOMES:
Dyspnea (breathlessness) | Assessed every 2-minutes until completion of the exercise trial; anticipating ~10-14 minute tests
  Particpants will rate their perceived dyspnea (breathlessness) using the modified Borg 0-10 scale (0 - No breathlessness; 10 - Maximal breathlessness)
Pulmonary artery systolic pressure | Assessed for five consecutive cardiac cycles and are measured in triplicate during the cardiac ultrasound trial. This will be completed within 4 weeks of enrollment in the study.
  Pulmonary artery systolic pressure will be assessed at rest and during exercise
Emphysema severity score | Emphysema severity score assessed by computed tomography. This will be completed within 4 weeks of enrollment in the study.
  Emphysema severity score assessed by computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Sciences Building, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No